CLINICAL TRIAL: NCT00006107
Title: Taxotere Plus Concurrent Concomitant Boost Radiotherapy For Squamous Cell Cancer of the Head and Neck (TAXT-XRT)
Brief Title: Chemotherapy and Radiation Therapy in Treating Patients With Stage III or Stage IV Head and Neck Cancer
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Dana-Farber Cancer Institute (Other)
Collaborators: National Cancer Institute (NCI) (NIH)
Responsible Party: Principal Investigator, Roy B. Tishler, MD, Principal Investigator, Dana-Farber Cancer Institute
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 99-274; P30CA006516 (NIH); NCI-G00-1833
Record Dates: First submitted 2000-08-03; First posted 2003-01-27 (Estimated); Last update posted 2017-06-16 (Actual); Status verified 2017-06

CONDITIONS: Head and Neck Cancer
Keywords: recurrent metastatic squamous neck cancer with occult primary; metastatic squamous neck cancer with occult primary squamous cell carcinoma; stage III squamous cell carcinoma of the lip and oral cavity; stage IV squamous cell carcinoma of the lip and oral cavity; recurrent squamous cell carcinoma of the lip and oral cavity; stage III squamous cell carcinoma of the oropharynx; stage IV squamous cell carcinoma of the oropharynx; recurrent squamous cell carcinoma of the oropharynx; stage III squamous cell carcinoma of the nasopharynx; stage IV squamous cell carcinoma of the nasopharynx; recurrent squamous cell carcinoma of the nasopharynx; stage III squamous cell carcinoma of the hypopharynx; stage IV squamous cell carcinoma of the hypopharynx; recurrent squamous cell carcinoma of the hypopharynx; stage III squamous cell carcinoma of the larynx; stage IV squamous cell carcinoma of the larynx; recurrent squamous cell carcinoma of the larynx; stage III squamous cell carcinoma of the paranasal sinus and nasal cavity; stage IV squamous cell carcinoma of the paranasal sinus and nasal cavity; recurrent squamous cell carcinoma of the paranasal sinus and nasal cavity; recurrent salivary gland cancer; stage III salivary gland cancer; stage IV salivary gland cancer; salivary gland squamous cell carcinoma; recurrent lymphoepithelioma of the nasopharynx; recurrent lymphoepithelioma of the oropharynx; stage III lymphoepithelioma of the nasopharynx; stage III lymphoepithelioma of the oropharynx; stage IV lymphoepithelioma of the nasopharynx; stage IV lymphoepithelioma of the oropharynx
MeSH Terms: conditions — Head and Neck Neoplasms; Squamous Cell Carcinoma of Head and Neck; Salivary Gland Neoplasms | interventions — Docetaxel; Surgical Procedures, Operative; Radiotherapy

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (1):
- Taxotere (Experimental): * Taxotere: (1 hour infusion once a week for four weeks)
  * Radiation Therapy (5 days/week for 6-7 weeks)
  * Surgery (if required) 14 -12 weeks after radiotherapy
  * Follow-up
  Interventions: Drug: Taxotere; Procedure: Surgery; Radiation: radiation therapy

INTERVENTIONS:
Drug: Taxotere
  Other Names: Docetaxel
Procedure: Surgery
Radiation: radiation therapy

SUMMARY:
Phase I trial to study the effectiveness of docetaxel plus radiation therapy in treating patients who have stage III or stage IV head and neck cancer.

DETAILED DESCRIPTION:
OBJECTIVES:

* Determine the maximum tolerated dose of docetaxel when administered with concurrent boost radiotherapy in patients with advanced squamous cell carcinoma of the head and neck previously treated with induction chemotherapy.
* Determine the toxicity of this treatment regimen in this patient population.
* Determine the efficacy of this treatment regimen in these patients.

OUTLINE: This is a dose escalation study of docetaxel.

Patients receive docetaxel IV over 1 hour weekly for 4 weeks. Patients also undergo hyperfractionated radiotherapy daily, 5 days a week, for 4 weeks followed by radiotherapy alone twice daily for 2 weeks.

Upon completion of chemoradiotherapy, patients not achieving complete response to induction chemotherapy undergo neck surgical dissection at 4-12 weeks following completion of radiotherapy.

Cohorts of 3-5 patients receive escalating doses of docetaxel until the maximum tolerated dose (MTD) is reached. The MTD is the dose preceding that at which 2 of 3 or 2 of 5 patients experience dose limiting toxicity. Additional patients are treated at the MTD.

Patients are followed monthly for 1 year, and then annually thereafter.

PROJECTED ACCRUAL: A total of 18-25 patients will be accrued for this study.

ELIGIBILITY:
Inclusion Criteria:

* Pathology:

  -- Histologic documentation of squamous cell carcinoma of the head and neck or its variants (lymphoepithelioma, undifferentiated epidermoid carcinoma, etc.).
* Stage:

  -- Patients will be entered on this protocol after initial induction therapy, if, prior to the induction regimen, they were previously untreated Stage III or IV (MO) SCCHN. Evaluable disease during induction therapy is required.
  * Required Prior Therapy: Patients entered on this protocol will have received platinum/FUra based induction chemotherapy. They may have received a taxane as part of this plan.
  * Patients treated with induction are eligible provided that they receive no more than 3 cycles of chemotherapy, but at least one cycle of chemotherapy, and are less then 7 weeks from the start of last cycle of induction therapy.
* Other Malignancies:

  * Patients with previous head and neck cancer are ineligible, except patients who were treated with surgery as the sole modality ≥2 years prior to study entry.
  * Patients with concurrent malignancy of any site, except limited basal cell carcinoma or squamous cell carcinoma of the skin or carcinoma in situ of the cervix are ineligible.
  * Patients with any non-SCCHN malignancy within 3 years of study entry, except curatively treated basal cell carcinoma or squamous cell carcinoma of the skin or carcinoma in situ of the cervix are ineligible.
* Other Prior Therapy:

  * Patients treated with induction therapy
  * Hormonally treated patients are eligible.
* Performance: Patients must meet the following performance criteria:

  * Performance status: ≤2 (ECOG) Complete recovery from previous diagnostic or therapeutic procedures is required.
  * Nutritional Status: Adequate and nutritionally balanced enteral intake ≥ 1,800 kcal/day).
  * A PEG is required prior to initiation of radiation.
  * Age: ≥18 years
  * Life Expectancy: Longer than 3 months.
  * Women of child bearing potential must not be pregnant by history or lactating at the time of entry on this protocol and men and women of child bearing potential must be requested to use an accepted and effective method of birth control during therapy.
* Organ Function: Biochemical and hematological parameters (obtained within 2 weeks of study entry) as follows:

  * Hepatic: SGOT < 1.5 x ULN and Alkaline Phosphatase < 2.5 x ULN for entry. Total Bilirubin = WNL and SGOT must be ≤ 2 x ULN as an isolated value. SGPT ≤ 2.5 x ULN
  * Hematologic: WBC ≥ 3,000/mm3 or a normal absolute neutrophil count (ANC) ≥ 1000; Platelet count ≥ 100,000/mm3 Hemoglobin ≥ 10 gm/d1 (transfusion to bring the hemoglobin to or above this level is permitted if clinically indicated, however, transfusions should not be used solely in order to meet eligibility criteria).
* Neurologic: Peripheral neuropathy of any etiology must not exceed grade 2.
* Other: Lack of other serious illness or medical condition
* Informed consent:

  -- Patients must give written informed consent.
* Follow-up:

  * All patients must be available for monthly evaluation and re-staging by the physicians from the Head and Neck Cancer Clinic while on therapy.

Exclusion Criteria:

* Pathology:

  -- Patients with previous head and neck cancer are ineligible, except patients who were treated with surgery as the sole modality ≥ 2 years prior to study entry.
* Other Malignancies:

  * Patients with concurrent malignancy of any site, except limited basal cell carcinoma or squamous cell carcinoma of the skin or carcinoma in situ of the cervix are ineligible.
  * Patients with any non-SCCHN malignancy within 3 years of study entry, except curatively treated basal cell carcinoma or squamous cell carcinoma of the skin or carcinoma in situ of the cervix are ineligible.
* Other Prior Therapy:

  * Patients who were previously treated with radiotherapy for SCCHN are not eligible.
  * Patients treated with any form of prior chemotherapy, other than induction therapy within the last 5 years are not eligible
* Performance:

  * Nutritional Status: Patients requiring intravenous alimentation as primary source of calories are excluded from this study.
  * Patients with persistent diarrhea are ineligible.
* Organ Function:

  -- Neurologic: Peripheral neuropathy of any etiology must not exceed grade 2.

  -- Cardiovascular/Pulmonary: No acute cardiac dysrhythmias or unstable cardiac condition such as angina.
* Follow-up:

  * Patients with a history of severe hypersensitivity reaction to Taxotere or other drugs formulated with polysorbate 80 will be excluded.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 31 (Actual)
Dates: Start 2000-07-14 (Actual); Primary Completion 2003-07-17 (Actual); Study Completion 2004-07-03 (Actual)

PRIMARY OUTCOMES:
MTD of Taxotere | 8 Weeks
Dose Limiting Toxicity | 8 Weeks

SECONDARY OUTCOMES:
Overall Response Rate | 4-12 weeks post chemo/radiation therapy
Tumor Resistance Predictors | Up to 1 year post chemo/radiation therapy
  Tumor Biopsies and tissues

CONTACTS AND LOCATIONS:
Overall Officials: Roy B. Tishler, MD, PhD, Principal Investigator — Dana-Farber Cancer Institute
Locations (2):
- United States (2):
  - Massachusetts General Hospital, Boston, Massachusetts
  - Dana Farber Cancer Institute, Boston, Massachusetts

IPD SHARING:
Plan to Share IPD: No